CLINICAL TRIAL: NCT03785977
Title: A Prospective Comparison of the Airway Deadspace Associated With the Air-Q® and Endotracheal Tube Using Volumetric Capnography in Young Children
Brief Title: Airway Deadspace in Children: Air-Q Versus Endotracheal Tube
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00055260
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Airway Deadspace
Keywords: Ventilation; pediatrics; airway management; respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Air-Q 5-9kg: Participants weighing 5-9kg may be chosen to wear the Air-Q device.
- Air-Q 10-14kg: Participants weighing 10-14kg may be chosen to wear the Air-Q device.
- Air-Q 15-20kg: Participants weighing 15-20kg may be chosen to wear the Air-Q device.
- ETT 5-9kg: Participants weighing 5-9kg may be chosen to wear the ETT device.
- ETT 10-14kg: Participants weighing 10-14kg may be chosen to wear the ETT device.
- ETT 15-20kg: Participants weighing 15-20kg may be chosen to wear the ETT device.

SUMMARY:
The objective of this study will be to measure the airway deadspace associated with use of appropriately sized an AirQ, a commonly used supraglottic airway in young children weighing between 5 and 20 kg and compare that to the airway deadspace associated with use of an endotracheal tube (ETT) in similarly sized children undergoing controlled ventilation.

DETAILED DESCRIPTION:
There is an increasing interest in the use of supraglottic airway devices in progressively younger and younger patients. One issue that has not been well evaluated is the contribution of these devices to airway dead space in young children and infants. Volumetric capnography is the only non-invasive technology available at the current time to evaluate airway deadspace. Volumetric capnography essentially monitors the flow of CO2 over time and from the expired waveform one can determine different respiratory parameters including dead space. This is clinically important in young children as the clinician begins to evaluate whether or not to use an endotracheal tube or supraglottic airway in these patients. To perform this investigation the study team will use volumetric capnography to examine the airway dead space associated with these devices during and elective general surgery and urologic procedures in healthy children between the ages of 0 and 6 years of age (roughly 5-20 kg).

Participants in the study will be given ETT or Air-Q as an intervention, but the investigator does not assign specific interventions to the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 3 months and 6 years of age weighing between 5 and 20 kg
* Patient presenting outpatient urologic or general surgery

Exclusion Criteria:

* History of difficult airway/intubation
* Patients suspected to have a difficult airway.
* Morbid obesity BMI >39
* Emergency status of surgery
* Patients exposed to second hand smoke
* Patients with Asthma
* Patients with a URI symptom such as nasal drainage, cough, or fever within 7 days of the date of surgery
* History of Prematurity

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: To perform this investigation we will use volumetric capnography to examine the airway dead space associated with these devices during and elective general surgery and urologic procedures in healthy children between the ages of 0 and 5 years of age (roughly 5-20 kg).
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Mean Value of Airway Dead Space | 10 minutes
  A mean value observed over the first 10 minutes following placement of the ETT or the AirQ at the beginning of the case will be recorded.

SECONDARY OUTCOMES:
Lung Compliance measured by Respironics NM3 respiratory monitors | 10 minutes
  The values of lung compliance will be collected and reported.
Airway Resistance measured by Respironics NM3 respiratory monitors | 10 minutes
  The value of resistance to flow in the airways will be collected and reported
Volume of Carbon Dioxide Associated with the Devices | 10 minutes
  The volume of carbon dioxide associated with the devices will be recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Templeton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Micaglio M, Bonato R, De Nardin M, Parotto M, Trevisanuto D, Zanardo V, Doglioni N, Ori C. Prospective, randomized comparison of ProSeal and Classic laryngeal mask airways in anaesthetized neonates and infants. Br J Anaesth. 2009 Aug;103(2):263-7. doi: 10.1093/bja/aep106. Epub 2009 May 19. PMID 19454544
- [Background] Templeton TW, Hoke LK, Templeton LB, Ririe DG, Rose DM, Bryan YF. A comparison of 3 ventilation strategies in children younger than 1 year using a Proseal laryngeal mask airway: a randomized controlled trial. J Clin Anesth. 2016 Dec;35:502-508. doi: 10.1016/j.jclinane.2016.07.042. Epub 2016 Oct 19. PMID 27871584
- [Background] Garcia-Fernandez J, Tusman G, Suarez-Sipmann F, Llorens J, Soro M, Belda JF. Programming pressure support ventilation in pediatric patients in ambulatory surgery with a laryngeal mask airway. Anesth Analg. 2007 Dec;105(6):1585-91, table of contents. doi: 10.1213/01.ane.0000287674.64086.f1. PMID 18042854
- [Background] Drake-Brockman TF, Ramgolam A, Zhang G, Hall GL, von Ungern-Sternberg BS. The effect of endotracheal tubes versus laryngeal mask airways on perioperative respiratory adverse events in infants: a randomised controlled trial. Lancet. 2017 Feb 18;389(10070):701-708. doi: 10.1016/S0140-6736(16)31719-6. Epub 2017 Jan 18. PMID 28108038
- [Background] Casati A, Fanelli G, Torri G. Physiological dead space/tidal volume ratio during face mask, laryngeal mask, and cuffed oropharyngeal airway spontaneous ventilation. J Clin Anesth. 1998 Dec;10(8):652-5. doi: 10.1016/s0952-8180(98)00108-1. PMID 9873966
- [Background] Templeton TW, Goenaga-Diaz EJ, Templeton LB, Ririe DG. An in vitro analysis of the dead space in 5 supraglottic airway devices intended for use in small children and infants. Paediatr Anaesth. 2018 Jun;28(6):570-572. doi: 10.1111/pan.13382. No abstract available. PMID 29878544
- [Background] Templeton TW, Hoke LK, Yaung J, Aschenbrenner CA, Rose DM, Templeton LB, Bryan YF. Comparing 3 ventilation modalities by measuring several respiratory parameters using the ProSeal laryngeal mask airway in children. J Clin Anesth. 2016 Nov;34:272-8. doi: 10.1016/j.jclinane.2016.04.031. Epub 2016 May 15. PMID 27687391
- [Background] Al-Subu A, Jooste E, Hornik CP, Fleming GA, Cheifetz IM, Ofori-Amanfo G. Correlation between minute carbon dioxide elimination and pulmonary blood flow in single-ventricle patients after stage 1 palliation and 2-ventricle patients with intracardiac shunts: A pilot study. Paediatr Anaesth. 2018 Jul;28(7):618-624. doi: 10.1111/pan.13423. PMID 30133920
- [Background] Ream RS, Schreiner MS, Neff JD, McRae KM, Jawad AF, Scherer PW, Neufeld GR. Volumetric capnography in children. Influence of growth on the alveolar plateau slope. Anesthesiology. 1995 Jan;82(1):64-73. doi: 10.1097/00000542-199501000-00010. PMID 7832337